CLINICAL TRIAL: NCT05843188
Title: A Phase II Study of 5-FU, Irinotecan, Bevacizumab and Hydroxychloroquine in Drug-Tolerant Persister (DTP)-Selected Patients With Metastatic Colorectal Cancer
Brief Title: Study of Hydroxychloroquine With FOLFIRI and Bevacizumab in DTP-high Metastatic Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Targeting DTP in mCRC; 22-5689 (Other: University Health Network)
Record Dates: First submitted 2023-03-29; First posted 2023-05-06 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Hydroxychloroquine; Irinotecan; Leucovorin; Fluorouracil; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High DTP-signature (Experimental): Take HCQ, 400 mg by mouth, twice daily. Receive FOLFIRI+bevacizumab (irinotecan 180 mg/m2, leucovorin 400 mg/m2, 5-FU 2400 mg/m2 over 46 - 48 hours, bevacizumab 5 mg/kg), intravenously, every 2 weeks
  Interventions: Drug: Hydroxychloroquine; Drug: Irinotecan; Drug: Leucovorin; Drug: Fluorouracil; Drug: Bevacizumab
- Low DTP-signature (Active Comparator): Receive FOLFIRI+bevacizumab (irinotecan 180 mg/m2, leucovorin 400 mg/m2, 5-FU 2400 mg/m2 over 46 - 48 hours, bevacizumab 5 mg/kg), intravenously, every 2 weeks
  Interventions: Drug: Irinotecan; Drug: Leucovorin; Drug: Fluorouracil; Drug: Bevacizumab

INTERVENTIONS:
Drug: Hydroxychloroquine — Anti-Inflammatory - antimalarial - aminoquinolines
  Arms: High DTP-signature
Drug: Irinotecan — Antineoplastic agent
Drug: Leucovorin — Folic acid derivative
  Other Names: Folinic acid
Drug: Fluorouracil — Antineoplastic agent
  Other Names: 5-FU
Drug: Bevacizumab — Antineoplastic agent

SUMMARY:
This is a two arm, 2-center, Phase II, study of 5-FU, irinotecan, bevacizumab (FOLFIRI-beva) and hydroxychloroquine (HCQ) in patients with previously untreated metastatic colorectal cancer (mCRC).

Up to 155 patients will be screened for DTP-signature and up to 31 evaluable patients who are determined to be DTP-signature high will be treated with FOLFIRI-beva and HCQ.

Patients will continue to receive treatments until evidence of disease progression, intolerable side effects, withdrawal of consent or death.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal cancer, not amenable to curative resection.
* Microsatellite stable/mismatch repair proficient (MSS/pMMR) colorectal cancer.
* No prior systemic therapy for metastatic disease.
* Evaluable disease based on RECIST 1.1 criteria.
* Adequate hematological, hepatic and renal functions
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-1.
* Estimated life expectancy of > 6 months.
* Negative pregnancy test for female patients with child-bearing potential.
* No history of retinal disorder.
* No history of glucose-6-phosphate dehydrogenase deficiency (G6PD) .
* Considered to be DTP-signature high to receive HCQ treatment

Exclusion Criteria:

* Women who are pregnant or nursing.
* Have received radiotherapy, chemotherapy, biological therapy, or investigational treatment less than four weeks (six weeks for nitrosoureas or mitomycin C) prior to first dose of FOLFIRI-beva or have not recovered from all acute toxicities from prior treatments to grade 1 or less, with the exception of alopecia and those deemed not to affect safety assessment.
* Have concurrent malignancy with exception of malignancy that was treated curatively and without evidence of recurrence within 3 years of study enrollment, or fully resected basal or squamous cell skin cancer and any carcinoma in situ which are considered to be of low risk of recurrence.
* Have had major surgery within 28 days of study enrollment. Placement of a venous access device within 28 days of starting therapy is allowed.
* Have any medical condition that would impair the administration of oral agents including significant bowel resection, inflammatory bowel disease or uncontrolled nausea or vomiting.
* Known central nervous system metastasis. Patients with history of central nervous system metastases are eligible if they are clinically and radiographically stable for at least 3 months and not taking steroids or anticonvulsants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2026-04-24 (Estimated); Study Completion 2026-10-24 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Start of study treatment to end of study, up to 48 months.
  Percentage of participants who have a partial response or complete response to study treatment.

SECONDARY OUTCOMES:
Progression-free survival | Start of study treatment to time of disease progression, up to 48 months.
  Average length of time that participants' diseases do not worsen.
Overall survival | Start of study treatment to time of death, up to 48 months.
  Average length of time that participants are alive.
Incidences and severity of adverse events | Start of study treatment to end of study, up to 48 months.
  Number of adverse events per grade

CONTACTS AND LOCATIONS:
Overall Officials: Eric Chen, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (2):
- Canada (2):
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario